CLINICAL TRIAL: NCT07248956
Title: Neoadjuvant Chemotherapy Combined With Finotonlimab in the Treatment of Locally Advanced Hypopharyngeal Carcinoma: A Multicenter Randomized Controlled Study
Brief Title: Neoadjuvant Chemotherapy Combined With Finotonlimab in the Treatment of Locally Advanced Hypopharyngeal Carcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Eye & ENT Hospital of Fudan University (Other)
Responsible Party: Principal Investigator, Ming Zhang, Principal Investigator, Eye & ENT Hospital of Fudan University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SOAR-HP
Record Dates: First submitted 2025-11-18; First posted 2025-11-25 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Hypopharyngeal Carcinoma
Keywords: PD-1 inhibitor; neoadjuvant therapy; locally advanced
MeSH Terms: conditions — Hypopharyngeal Neoplasms | interventions — Albumin-Bound Paclitaxel; 130-nm albumin-bound paclitaxel; Cisplatin; Surgical Procedures, Operative; Chemoradiotherapy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- neoadjuvant therapy followed by surgery and (C)RT group (Experimental): Patients initially receive immunotherapy with Finolizumab and chemotherapy with albumin-bound paclitaxel and cisplatin. Patients with response of complete reaction (CR)/partial reaction (PR)≥50% after neoadjuvant chemotherapy then receive surgery, followed by postoperative radiotherapy or chemoradiotherapy.
  Interventions: Drug: Finolizumab; Drug: Albumin-Bound Paclitaxel /nab-Paclitaxel; Drug: Cisplatin; Procedure: Surgery with postoperative radiotherapy or chemoradiotherapy.
- neoadjuvant therapy followed by CCRT group (Active Comparator): Patients initially receive immunotherapy with Finolizumab and chemotherapy with albumin-bound paclitaxel and cisplatin. Patients with response of complete reaction (CR)/partial reaction (PR)≥50% after neoadjuvant chemotherapy then receive definitive radiotherapy with concurrent cisplatin-based chemotherapy.
  Interventions: Drug: Finolizumab; Drug: Albumin-Bound Paclitaxel /nab-Paclitaxel; Drug: Cisplatin; Radiation: Definitive radiotherapy

INTERVENTIONS:
Drug: Finolizumab — 200mg every 3 weeks (q3w) for 2 cycles.
Drug: Albumin-Bound Paclitaxel /nab-Paclitaxel — 260mg/m², day 1, every 3 weeks (q3w) for 2 cycles.
Drug: Cisplatin — 25mg/m², days 1-3, every 3 weeks (q3w) for 2 cycles.
Radiation: Definitive radiotherapy — Definitive radiotherapy (68-70Gy) with concurrent cisplatin-based chemotherapy (25mg/m², days 1-3, every 3 weeks)
  Arms: neoadjuvant therapy followed by CCRT group
Procedure: Surgery with postoperative radiotherapy or chemoradiotherapy. — surgery with postoperative radiotherapy or chemoradiotherapy.
  Arms: neoadjuvant therapy followed by surgery and (C)RT group

SUMMARY:
This is a multi-center, randomized controlled, prospective clinical study.

DETAILED DESCRIPTION:
The early symptoms of hypopharyngeal cancer are often inconspicuous, with approximately 70% of patients clinically diagnosed at an advanced stage. With the emergence of immunotherapy, immune therapies such as PD-1 inhibitors combined with induction chemotherapy have been widely explored in various tumor types. Currently, there is a lack of large-scale real-world studies on the efficacy and safety of treatment options for patients with locally advanced hypopharyngeal cancer who respond well to neoadjuvant therapy. This study aims to employ neoadjuvant chemotherapy combined with immunotherapy for locally advanced hypopharyngeal cancer and explore the effectiveness and safety of different subsequent treatment options for patients assessed as achieving a major partial response (PR ≥50%).

ELIGIBILITY:
Inclusion Criteria:

1. Willingness to provide written informed consent;
2. Age ≥18 and ≤75 years;
3. Treatment-naïve for malignant disease;
4. Resectable stage III-IVA hypopharyngeal carcinoma with response of PR ≥ 50% after neoadjuvant therapy according to RECIST 1.1 ;
5. ECOG performance status 0-2.

Exclusion Criteria:

1. Pregnancy or breastfeeding status;
2. Hypersensitivity to sintilimab, nab-paclitaxel, or their formulation components;
3. Poorly controlled cardiovascular conditions or other diseases;
4. Active or documented history of autoimmune diseases requiring systemic treatment;
5. Synchronous or metachronous malignancies;
6. Other conditions deemed ineligible for the study by investigators.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Estimated)
Dates: Start 2025-12-22 (Actual); Primary Completion 2027-11-30 (Estimated); Study Completion 2029-12-30 (Estimated)

PRIMARY OUTCOMES:
Event-free survival (EFS) | 2 years
  Duration from treatment initiation until the first occurrence of any of the following events: disease progression precluding surgical intervention, local or distant recurrence, death from any cause, etc.

SECONDARY OUTCOMES:
Overall Survival (OS) | 2 years
  Duration from the date of tumor treatment initiation to the date of first documented death from any cause or the last follow-up date.
Locoregional Control Rate (LRFS) | 2 years
  Duration from the date of tumor treatment initiation to the date of first documented locoregional recurrence, death from any cause, or the last follow-up date.
Laryngeal Preservation Rate | 2 years
  The proportion of patients who successfully retain laryngx function after treatment.
Major Pathological Response Rate (MPR) | 2 years
  The presence of ≤10% viable invasive squamous cell carcinoma in the resected primary tumor and neck lymph nodes.
Adverse events | 2 years
  Acute treatment-related toxicities were evaluated using CTCAE v5.0 (Common Terminology Criteria for Adverse Events, Version 5.0), with patient counts reported for each AE category.
  Late radiation toxicities were assessed per the RTOG (Radiation Therapy Oncology Group) grading criteria, with both patient numbers and incidence rates documented.

CONTACTS AND LOCATIONS:
Overall Officials: Ming Zhang, PhD, Principal Investigator — Eye & ENT Hospital, Fudan University
Locations (7):
- China (7):
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - Shandong Provincial ENT Hospital, Jinan, Shandong
  - Beijing Tongren Hospital, Capital Medical University, Beijing
  - Cancer Hospital Chinese Academy of Medical Sciences, Beijing
  - Eye & ENT Hospital, Fudan University, Shanghai
  - Zhongshan Hospital of Fudan University, Shanghai
  - Tianjin Medical University Cancer Institute & Hospital, Tianjin

IPD SHARING:
Plan to Share IPD: No